CLINICAL TRIAL: NCT03028870
Title: A Phase 2a, Multicenter, Randomized, Double-blind, Placebo-controlled and Active-controlled, Parallel-group Study Evaluating the Analgesic Efficacy and Safety of V120083 in Subjects With Moderate to Severe Chronic Pain Due to Osteoarthritis of the Knee
Brief Title: A Study to Evaluate the Analgesic Efficacy and Safety of V120083 in Subjects With Osteoarthritis (OA) of the Knee
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Purdue Pharma LP (Industry)
Collaborators: Shionogi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VAN2001
Record Dates: First submitted 2017-01-19; First posted 2017-01-23 (Estimated); Results first posted 2018-11-15 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-01

CONDITIONS: Osteo Arthritis Knee
Keywords: Osteoarthritis; Pain; Osteoarthritis Knee
MeSH Terms: conditions — Osteoarthritis; Pain; Osteoarthritis, Knee | interventions — Naproxen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- V120083 30 mg (Experimental): V120083 30-mg capsules taken orally twice daily
  Interventions: Drug: V120083; Drug: Placebo
- V120083 60 mg (Experimental): V120083 60-mg (2 x 30 mg) capsules taken orally twice daily
  Interventions: Drug: V120083; Drug: Placebo
- Naproxen (Active Comparator): Naproxen 500-mg capsules taken orally twice daily
  Interventions: Drug: Naproxen; Drug: Placebo
- Placebo (Placebo Comparator): Capsules to match V120083 and/or naproxen taken orally twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: V120083 — Capsules
  Arms: V120083 30 mg; V120083 60 mg
Drug: Naproxen — Capsules
  Arms: Naproxen
Drug: Placebo — Capsules to match V120083 and/or naproxen

SUMMARY:
The purpose of this study is to evaluate the analgesic efficacy of V120083 twice daily compared to placebo in subjects with moderate to severe chronic pain due to OA of the knee.

ELIGIBILITY:
Key Inclusion Criteria Include:

1. Males and females ≥ 40 and ≤ 80 years of age with moderate to severe chronic OA pain of the knee (lasting several hours daily) as their predominant pain condition for at least 6 months prior to screening
2. Diagnostic criteria for primary pain condition (American College of Rheumatology [ACR] clinical and radiographic criteria):

   * At least 1 of the following in addition to knee pain: age > 50, morning stiffness < 30 minutes, crepitus on active motion, and
   * Kellgren-Lawrence (K-L) grade 2 or 3 radiographic evidence at the screening visit as determined by a local radiologist or rheumatologist. If a radiograph is not available, one must be taken and the diagnostic criteria must be confirmed before randomization.
3. Subjects whose OA pain of the index knee is not adequately treated prior to the screening visit:

   * Subjects must have a self-reported average pain intensity rating of moderate or severe on a verbal rating scale (ie, none, mild, moderate, and severe) over the 7 days prior to the screening visit
4. The subjects must have "average pain over the last 24 hours" scores ≥ 4 and ≤ 9 on an 11-point numerical rating scale (NRS) for the index knee on ≥ 3 consecutive days during the pain assessment period and come in for randomization within 96 hours after the latest qualifying pain score entry
5. Subjects who are willing and able to stop taking any/all analgesic medications, including over-the-counter pain medications, opioids, marijuana, and topical analgesics for OA pain for the duration of the study, with the exception of study-specific rescue medication.

Key Exclusion Criteria Include:

1. Subjects with radiographic evidence of OA with K-L grade 0,1 or 4
2. Subjects with chronic pain conditions other than OA of the knee as their predominant pain condition, including gout, pseudogout, psoriatic arthritis, active Lyme disease, rheumatoid arthritis or any other inflammatory arthritis, fibromyalgia, neuropathic pain conditions, bursitis, or acute injury or signs of active infection in the target pain area
3. Subjects scheduled for surgical interventions of the disease site or any other major surgery during the study conduct period
4. Subjects with a history of a prior joint replacement of the index knee
5. Subjects who have had arthroscopy on either knee or hip within 6 months of entering the study, or open surgery on either knee or hip within 12 months of entering the study
6. Subjects with a history of significant trauma to a knee, hip or shoulder within the previous year
7. Subjects who have significant pain, other than or more than knee pain, including significant hip, back pain, that may confound the analgesic efficacy assessments of this study.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 291 (Actual)
Dates: Start 2017-03-14 (Actual); Primary Completion 2017-11-10 (Actual); Study Completion 2017-11-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (30):
- United States (30):
  - Alabama Clinical Therapeutics, LLC, Birmingham, Alabama
  - Terence T. Hart, MD, Tuscumbia, Alabama
  - Providence Clinical Research, North Hollywood, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Artemis Institute for Clinical Research, San Marcos, California
  - Future Care Solution, LLC, Miami, Florida
  - New Horizon Research Center, Miami, Florida
  - Sensible Healthcare, LLC, Ocoee, Florida
  - Omega Research Consultants, LLC, Orlando, Florida
  - Clinical Research of West Florida, Inc., Tampa, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Buynak Clinical Research, P.C., Valparaiso, Indiana
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - St. Louis Center for Clinical Research, St Louis, Missouri
  - St. Louis Clinical Trials, LC, St Louis, Missouri
  - Sundance Clinical Research, LLC, St Louis, Missouri
  - Hassman Research Institute, Berlin, New Jersey
  - Drug Trials America, Hartsdale, New York
  - Montefiore Medical Center, The Bronx, New York
  - Medication Management, LLC, Greensboro, North Carolina
  - Research Institute of the Carolinas of Piedmont Healthcare, PA, Mooresville, North Carolina
  - Burke Primary Care, Morganton, North Carolina
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - New Horizons Clinical Research, Cincinnati, Ohio
  - Providence Health Partners - Center for Clinical Research, Dayton, Ohio
  - Omega Medical Research, Warwick, Rhode Island
  - Mountain View Clinical Research, Inc., Greer, South Carolina
  - FutureSearch Trials of Neurology, Austin, Texas
  - Diagnostics Research Group, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject first visit: 14-Mar-2017; last subject last visit: 21-Nov-2017. Thirty-one investigative centers in the United States participated in the study.
Groups:
- V120083 30 mg: V120083 30 mg taken orally twice daily
- V120083 60 mg: V120083 60 mg taken orally twice daily
- Naproxen: Naproxen 500 mg taken orally twice daily
- Placebo: To match V120083 and/or naproxen taken orally twice daily
Period: Overall Study
Arm/Group | V120083 30 mg | V120083 60 mg | Naproxen | Placebo
Started | 74 | 67 | 76 | 74
Completed | 57 | 57 | 60 | 65
Not Completed | 17 | 10 | 16 | 9
Not completed — Adverse Event | 7 | 4 | 3 | 3
Not completed — Withdrawal by Subject | 1 | 1 | 1 | 2
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 3 | 0 | 0 | 0
Not completed — Administrative | 5 | 5 | 12 | 4

BASELINE CHARACTERISTICS:
Population: The safety population (N = 291) was the group of subjects who were randomized and received at least 1 dose of the double-blind study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | V120083 30 mg | V120083 60 mg | Naproxen | Placebo | Total
Number analyzed (Participants) | 74 | 67 | 76 | 74 | 291
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.9 (8.66) | 60.7 (8.62) | 59.8 (8.94) | 59.0 (8.97) | 60.1 (8.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 42 | 49 | 46 | 183
  Male | 28 | 25 | 27 | 28 | 108
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 51 | 48 | 61 | 54 | 214
  Black or African American | 19 | 18 | 14 | 19 | 70
  Asian | 2 | 1 | 0 | 1 | 4
  American Indian or Alaskan Native | 1 | 0 | 0 | 0 | 1
  Other | 1 | 0 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Daily "Average Pain Over the Last 24 Hours" Score at Week 4
Description: At week 4, subjects were asked to rate their pain on an 11-point numerical scale where 0 = no pain, 10 = pain as bad as you can imagine.
Time Frame: Week 4
Population: The full analysis population (FAP) (N = 291) was the group of subjects who were randomized and received at least 1 dose of the double-blind study drug, and had at least 1 efficacy assessment.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | V120083 30 mg | V120083 60 mg | Naproxen | Placebo
Number analyzed (Participants) | 74 | 67 | 76 | 74
score on a scale
  Baseline | 5.9 (0.20) | 5.9 (0.18) | 6.1 (0.16) | 5.9 (0.21)
  Week 4: number analyzed (Participants) | 72 | 65 | 76 | 73
  Week 4 | 4.2 (0.28) | 4.3 (0.28) | 3.6 (0.26) | 4.4 (0.29)

2. Secondary Outcome: Weekly Change From Baseline Score of "Average Pain Over the Last 24 Hours" From the mBPI-SF Pain Severity Subscale
Description: Subjects were asked to rate their pain on an 11-point numerical scale where 0 = no pain, 10 = pain as bad as you can imagine.
Time Frame: Weeks 1, 2 and 4
Population: The FAP (N=291) was the group of subjects who were randomized and received at least 1 dose of the double-blind study drug, and had at least 1 efficacy assessment.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | V120083 30 mg | V120083 60 mg | Naproxen | Placebo
Number analyzed (Participants) | 74 | 67 | 76 | 74
score on a scale
  Baseline | 6.242 (0.1530) | 6.431 (0.1408) | 6.469 (0.1426) | 6.543 (0.1497)
  Week 1 change from baseline: number analyzed (Participants) | 69 | 65 | 75 | 72
  Week 1 change from baseline | -0.920 (0.1721) | -0.860 (0.1405) | -1.655 (0.1789) | -0.977 (0.1569)
  Week 2 change from baseline: number analyzed (Participants) | 61 | 62 | 72 | 70
  Week 2 change from baseline | -1.653 (0.2087) | -1.336 (0.1998) | -2.255 (0.2443) | -1.593 (0.1979)
  Week 4 change from baseline: number analyzed (Participants) | 56 | 55 | 59 | 63
  Week 4 change from baseline | -1.959 (0.2553) | -1.803 (0.2957) | -2.741 (0.2898) | -1.952 (0.2667)

3. Secondary Outcome: Average Daily "Pain Right Now" Score Collected by e-Diary
Description: as for outcome 2
Time Frame: 4 Weeks
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | V120083 30 mg | V120083 60 mg | Naproxen | Placebo
Number analyzed (Participants) | 74 | 67 | 76 | 74
score on a scale
  Baseline: number analyzed (Participants) | 46 | 35 | 43 | 42
  Baseline | 6.104 (0.1851) | 6.737 (0.2076) | 6.590 (0.2223) | 6.481 (0.2587)
  Week 4: number analyzed (Participants) | 8 | 9 | 1 | 8
  Week 4 | 6.366 (0.6400) | 7.269 (0.2627) | 6.000 (NA) — Since only one subject reported a pain score, standard error was not calculated. | 5.833 (0.7318)

4. Secondary Outcome: Western Ontario and McMaster Osteoarthritis Index (WOMAC) - Pain Subscale
Description: The pain subscale consisted of 5 items: walking; stair climbing; nocturnal; at rest; weight bearing. The score for each item ranged from 0 (none) to 4 (extreme). The pain subscale score was obtained by adding the responses to the 5 items which could range from 0 to 20.
Time Frame: 4 Weeks
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | V120083 30 mg | V120083 60 mg | Naproxen | Placebo
Number analyzed (Participants) | 74 | 67 | 76 | 74
score on a scale
  Baseline | 10.2 (0.40) | 9.6 (0.34) | 9.9 (0.34) | 10.1 (0.38)
  Week 4: number analyzed (Participants) | 72 | 65 | 76 | 73
  Week 4 | 7.0 (0.50) | 7.2 (0.48) | 5.5 (0.41) | 6.8 (0.46)

5. Secondary Outcome: Western Ontario and McMaster Osteoarthritis Index (WOMAC) - Stiffness Subscale
Description: The stiffness subscale consisted of 2 items; morning stiffness and stiffness occurring later in the day. The score for each item ranged from 0 (none) to 4 (extreme) and the stiffness subscale score was obtained by adding the responses to the 2 items which could range from 0 - 8.
Time Frame: 4 Weeks
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | V120083 30 mg | V120083 60 mg | Naproxen | Placebo
Number analyzed (Participants) | 74 | 67 | 76 | 74
score on a scale
  Baseline | 4.6 (0.17) | 4.5 (0.18) | 4.2 (0.17) | 4.5 (0.17)
  Week 4: number analyzed (Participants) | 72 | 65 | 76 | 73
  Week 4 | 3.2 (0.20) | 3.3 (0.24) | 2.6 (0.19) | 3.1 (0.20)

6. Secondary Outcome: Western Ontario and McMaster Osteoarthritis Index (WOMAC) - Physical Function Subscale
Description: The physical function subscale consisted of 17 items: descending stairs; ascending stairs; rising from sitting; standing; bending to floor; walking on flat surface; getting into or out of car; going shopping; putting on socks; rising from bed; taking off socks; lying in bed; sitting; getting into or out of the bathtub; getting on or off the toilet; heavy domestic duties; light domestic duties. The score for each item ranged from 0 (none) to 4 (extreme) and the physical function subscale score was obtained by adding the responses to the 17 items which could range from 0 to 68.
Time Frame: 4 Weeks
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | V120083 30 mg | V120083 60 mg | Naproxen | Placebo
Number analyzed (Participants) | 74 | 67 | 76 | 74
score on a scale
  Baseline | 34.6 (1.23) | 34.8 (1.13) | 33.6 (1.19) | 35.1 (1.23)
  Week 4: number analyzed (Participants) | 72 | 65 | 76 | 73
  Week 4 | 25.6 (1.73) | 25.0 (1.79) | 18.7 (1.46) | 23.2 (1.64)

7. Secondary Outcome: Western Ontario and McMaster Osteoarthritis Index (WOMAC) - Total Score
Description: The total score of the WOMAC consisted of 24 items (5 items from the pain subscale, 2 items from the stiffness subscale, and 17 items from the physical function subscale). The total score was obtained by adding the scores from these 3 subscales and could range from 0 to 96.
Time Frame: 4 Weeks
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | V120083 30 mg | V120083 60 mg | Naproxen | Placebo
Number analyzed (Participants) | 74 | 67 | 76 | 74
score on a scale
  Baseline | 49.3 (1.67) | 48.9 (1.54) | 47.6 (1.55) | 49.6 (1.65)
  Week 4: number analyzed (Participants) | 72 | 65 | 76 | 73
  Week 4 | 35.8 (2.35) | 35.5 (2.45) | 26.8 (1.99) | 33.1 (2.25)

8. Secondary Outcome: Modified Brief Pain Inventory-Short Form (mBPI-SF) - Total Score (All Parts of 6 Questions)
Description: The mBPI-SF consists of 6 questions and is a self-administered questionnaire used to assess the severity of pain, and the interference of pain on daily functions. Subjects rated their severity of pain / interference of pain on a 0 (no pain / does not interfere) to 10 (as bad as you can imagine / completely interferes) numerical rating scale (NRS) The total score is the sum of all parts of the 6 questions and the total score range is 0 - 110.
Time Frame: 4 Weeks
Population: The FAP (N = 291) was the group of subjects who were randomized and received at least 1 dose of the double-blind study drug, and had at least 1 efficacy assessment.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | V120083 30 mg | V120083 60 mg | Naproxen | Placebo
Number analyzed (Participants) | 74 | 67 | 76 | 74
score on a scale
  Baseline | 55.5 (2.49) | 53.4 (2.30) | 56.0 (1.90) | 53.1 (2.50)
  Week 4: number analyzed (Participants) | 72 | 65 | 76 | 73
  Week 4 | 36.5 (2.97) | 35.3 (3.03) | 28.5 (2.51) | 35.7 (3.14)

9. Secondary Outcome: Modified Brief Pain Inventory-Short Form (mBPI-SF) Pain Severity Subscale Score
Description: The mBPI-SF is a self-administered questionnaire. The pain severity subscale of the mBPI-SF consists of 4 questions which ask the subjects to rate their severity of pain on a 0 to 10 NRS for worst pain, least pain, average pain, and current pain. The severity of pain was computed as the mean of questions 1-4. The mean severity of pain scores could range from 0 to 10.
Time Frame: 4 Weeks
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | V120083 30 mg | V120083 60 mg | Naproxen | Placebo
Number analyzed (Participants) | 74 | 67 | 76 | 74
score on a scale
  Baseline | 5.784 (0.2068) | 5.739 (0.1935) | 5.747 (0.1525) | 5.801 (0.1978)
  Week 4: number analyzed (Participants) | 72 | 65 | 76 | 73
  Week 4 | 4.139 (0.2840) | 4.135 (0.2771) | 3.510 (0.2543) | 4.308 (0.2900)

10. Secondary Outcome: Modified Brief Pain Inventory-Short Form (mBPI-SF) Pain Interference Subscale Score
Description: The mBPI-SF is a self-administered questionnaire. The pain interference subscale of the mBPI-SF consists of Question 6 which has 7 parts, all of which ask the subjects to rate the impact/interference of their pain on various functions, ie, general activity, mood, walking, normal work, relations with others, sleep, and enjoyment of life on a 0 to 10 NRS where 0 = does not interfere and 10 = completely interferes. The mean interference of pain scores could range from 0 to 10.
Time Frame: 4 Weeks
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | V120083 30 mg | V120083 60 mg | Naproxen | Placebo
Number analyzed (Participants) | 74 | 67 | 76 | 74
score on a scale
  Baseline | 4.618 (0.2717) | 4.348 (0.2573) | 4.718 (0.2186) | 4.278 (0.2721)
  Week 4: number analyzed (Participants) | 72 | 65 | 76 | 73
  Week 4 | 2.847 (0.2925) | 2.679 (0.2961) | 2.070 (0.2377) | 2.634 (0.3049)

11. Secondary Outcome: Responder to Treatment (Calculated as the Percentage Reduction of "Average Pain Over the Last 24 Hours") at Week 4
Description: A subject's response to treatment was defined as the percentage reduction from the baseline "average pain over the last 24 hours" score to the week 4 pain score from the mBPI-SF pain severity subscale. Responders were defined as having > 0 % reduction; non-responders were defined as having ≤ 0% reduction.
Time Frame: Week 4
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | V120083 30 mg | V120083 60 mg | Naproxen | Placebo
Number analyzed (Participants) | 74 | 67 | 76 | 74
Participants
  Responder - Yes | 46 | 42 | 57 | 42
  Responder - No | 28 | 25 | 19 | 32

12. Secondary Outcome: Medical Outcomes Study Short Form-36 (SF-36) - Physical Component Summary
Description: The SF-36 is a generic health survey with 36 items that measure functional health and well-being from the subject's perspective. The survey is summarized into 8 dimensions/scales: physical functioning (PF), role-physical (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role-emotional (RE), and mental health (MH).
  The Physical Component Summary is derived from 4 of the 8 health dimensions (aggregate of PF, RP, BP, and GH scales). The minimum score is 0 and the maximum score is 100. A higher score indicates a better health state.
Time Frame: 4 Weeks
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | V120083 30 mg | V120083 60 mg | Naproxen | Placebo
Number analyzed (Participants) | 74 | 67 | 76 | 74
score on a scale
  Baseline | 31.689 (0.9696) | 31.629 (0.9146) | 32.348 (1.0737) | 33.762 (1.0315)
  Week 4: number analyzed (Participants) | 72 | 65 | 76 | 73
  Week 4 | 35.515 (1.3008) | 36.277 (1.3584) | 39.372 (1.2486) | 37.826 (1.1440)

13. Secondary Outcome: Medical Outcomes Study Short Form-36 (SF-36) - Mental Component Summary
Description: The SF-36 is a generic health survey with 36 items that measure functional health and well-being from the subject's perspective. The survey is summarized into 8 dimensions/scales: physical functioning (PF), role-physical (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role-emotional (RE), and mental health (MH).
  The Mental Component Summary is derived from 4 of the 8 health dimensions,(aggregate of VT, SF, RE, and MH scales). The minimum score is 0 and the maximum score is 100. A higher score indicates a better health state.
Time Frame: 4 Weeks
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | V120083 30 mg | V120083 60 mg | Naproxen | Placebo
Number analyzed (Participants) | 74 | 67 | 76 | 74
score on a scale
  Baseline | 59.248 (0.9688) | 59.766 (1.1498) | 60.450 (0.8714) | 59.450 (1.0132)
  Week 4: number analyzed (Participants) | 72 | 65 | 76 | 73
  Week 4 | 59.596 (0.9615) | 59.560 (1.0785) | 60.921 (0.7819) | 60.948 (0.8835)

14. Secondary Outcome: European Quality of Life Scale - 5 Dimensions (EQ-5D-5L) to Measure Health Status
Description: EQ-5D-5L is a standardized generic measure of health status for clinical and economic appraisal based on a descriptive system that defines health in terms of 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. It includes a visual analogue scale (VAS) with scores ranging from 0 ("worst imaginable health state") to 100 ("best imaginable health state").
Time Frame: 4 Weeks
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | V120083 30 mg | V120083 60 mg | Naproxen | Placebo
Number analyzed (Participants) | 74 | 67 | 76 | 74
score on a scale
  Baseline VAS Score | 73.2 (2.04) | 72.9 (1.94) | 75.4 (1.88) | 74.6 (1.79)
  Week 4 VAS Score: number analyzed (Participants) | 72 | 65 | 76 | 73
  Week 4 VAS Score | 77.0 (2.17) | 77.4 (2.42) | 83.7 (1.37) | 81.4 (1.43)

15. Secondary Outcome: Patient Global Impression of Change (PGIC)
Description: The PGIC is an ordinal scale which assesses the change in overall status relative to the start of the study. The scale has only 1 item, which measures global change of overall status by the subject on a 7-point scale (very much improved, much improved, minimally improved, no change, minimally worse, much worse, very much worse), where 1 = very much improved and 7 = very much worse. The number of subjects responding "very much improved" and "much improved" was summarized by treatment group.
Time Frame: 4 Weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | V120083 30 mg | V120083 60 mg | Naproxen | Placebo
Number analyzed (Participants) | 74 | 67 | 76 | 74
Participants
  Total Subjects Completing PGIC | 72 | 65 | 76 | 72
  Subjects Responding 'Very Much' / 'Much' Improved | 25 | 27 | 38 | 18

16. Secondary Outcome: Supplemental Analgesic Medication Use
Description: The average daily number of tablets of supplemental pain medication used during the double-blind period was summarized by treatment group.
Time Frame: Up to 28 days
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Supplemental Analgesic Tablets
Arm/Group | V120083 30 mg | V120083 60 mg | Naproxen | Placebo
Number analyzed (Participants) | 38 | 35 | 34 | 40
Supplemental Analgesic Tablets | 0.779 (0.1471) | 0.686 (0.1187) | 0.378 (0.0712) | 0.670 (0.1205)

17. Secondary Outcome: Number of Participants With Treatment-emergent Suicidal Ideation and Behaviors Assessed by Columbia-Suicide Severity Rating Score (C-SSRS)
Description: Suicidality was monitored throughout the study using the C-SSRS. The C-SSRS involves a series of probing questions to inquire about possible suicidal thinking and behavior. The composite endpoints (Suicidal Ideation, Suicidal Behavior, Suicidal Ideation or Behavior) included subjects who experienced any one of the events at least once during treatment.
Time Frame: Baseline up to 4 Weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | V120083 30 mg | V120083 60 mg | Naproxen | Placebo
Number analyzed (Participants) | 74 | 67 | 76 | 74
Participants
  Suicidal ideation | 0 | 0 | 0 | 0
  Suicidal behavior | 0 | 0 | 0 | 0
  Suicidal ideation or behavior | 0 | 0 | 0 | 0
  Self-injurious behavior without suicidal intent | 0 | 0 | 0 | 0

18. Secondary Outcome: Change From Baseline to Week 4 in Hospital Anxiety and Depression Scale (HADS) Score
Description: Safety assessment to evaluate the impact of V120083 on mood (anxiety [HADS-A] and depression [HADS-D]). The score for each subscale ranges from 0 (no anxiety or depression) to 21, with a score of 11 or higher indicating the probable presence of the mood disorder.
Time Frame: Week 4
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | V120083 30 mg | V120083 60 mg | Naproxen | Placebo
Number analyzed (Participants) | 74 | 67 | 76 | 74
score on a scale
  Week 4 change from baseline - HADS-A: number analyzed (Participants) | 72 | 65 | 76 | 72
  Week 4 change from baseline - HADS-A | -0.5 (0.26) | -0.3 (0.26) | -0.4 (0.30) | -0.6 (0.35)
  Week 4 change from baseline - HADS-D: number analyzed (Participants) | 72 | 65 | 76 | 72
  Week 4 change from baseline - HADS-D | 0.3 (0.25) | 0.6 (0.31) | -0.2 (0.29) | -0.1 (0.30)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were reported from the start of study participation up to 5 weeks and from the start of study participation up to 30 days after last study drug dose for serious AEs.
Description: AEs were learned of through spontaneous reports and/or subject interview, or were observed during physical examinations or other safety assessments. Ongoing AEs were followed until resolution or for 30 days after last study drug dose. Serious AEs reported within 30 days after the subject's last study drug dose or through the last study visit (whichever was later), were followed until the event resolved or sequelae stabilized.
Arm/Group | V120083 30 mg | V120083 60 mg | Naproxen | Placebo
All-Cause Mortality (participants affected / at risk) | 0/74 | 0/67 | 0/76 | 0/74
Serious Adverse Events (participants affected / at risk) | 0/74 | 1/67 | 1/76 | 0/74
Other Adverse Events (participants affected / at risk) | 18/74 | 20/67 | 17/76 | 11/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | V120083 30 mg (N=74) | V120083 60 mg (N=67) | Naproxen (N=76) | Placebo (N=74)
Pyrexia (General disorders) | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Transaminases increased (Investigations) | 0 | 1 | 0 | 0
Delerium tremens (Psychiatric disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | V120083 30 mg (N=74) | V120083 60 mg (N=67) | Naproxen (N=76) | Placebo (N=74)
Nausea (Gastrointestinal disorders) | 5 | 5 | 9 | 4
Constipation (Gastrointestinal disorders) | 0 | 0 | 5 | 0
Decreased appetite (Metabolism and nutrition disorders) | 4 | 6 | 0 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 5 | 0 | 0
Dysgeusia (Nervous system disorders) | 13 | 13 | 7 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2017-02-16): https://cdn.clinicaltrials.gov/large-docs/70/NCT03028870/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-12): https://cdn.clinicaltrials.gov/large-docs/70/NCT03028870/SAP_001.pdf